CLINICAL TRIAL: NCT05624086
Title: Is There a Response of Hepatic Enzymes, Psychological Measures, and Sexual Dysfunction to Aerobic Exercise in Men With Sexual Dysfunction Complaint and Hepatitis C
Brief Title: Hepatic Enzymes, Psychological Measures, and Sexual Dysfunction Responses to Aerobic Exercise in Hepatitis-C Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004114
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Hepatitis C; Erectile Dysfunction
MeSH Terms: conditions — Hepatitis C; Erectile Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercised group (Experimental): In this group, Hepatitis-C Men With Sexual Dysfunction (erectile dysfunction) Complaint (n=23) will receive exercise-training sessions (one hour walking on treadmill, for 3 months, three walking sessions per the week)
  Interventions: Behavioral: exercise
- control group (No Intervention): in this group, Hepatitis-C Men With Sexual Dysfunction (erectile dysfunction) Complaint (n=23) will act as a control (waitlist) group that will receive no trainning

INTERVENTIONS:
Behavioral: exercise — Hepatitis-C Men With Sexual Dysfunction (erectile dysfunction) Complaint will receive exercise-training sessions (one hour walking on treadmill, for 3 months, three walking sessions per the week)
  Arms: Exercised group

SUMMARY:
Chronic hepatitis C virus (HCV) infection is a systematic disease that affects several aspects of patients' well-being, including physical, mental, social, and sexual quality of life. In recent years, this clinical trial aims to search the Response of Hepatic Enzymes, Psychological Measures, and Sexual Dysfunction to Aerobic Exercise in Hepatitis Men With Sexual Dysfunction Complaint

DETAILED DESCRIPTION:
Hepatitis Men With Sexual Dysfunction (erectile dysfunction) Complaint (n=46) will be randomized randomly to 23-men exercise-training (one hour walking on treadmill, for 3 months, three walking sessions per the week) hepatitis-C group or 23-men waiting-hepatitis-C group.

ELIGIBILITY:
Inclusion Criteria:

* men with hepatitis C men diagnosis
* men with sexual dysfunction (erectile dysfunction)

Exclusion Criteria:

* obesity , men with cardiac/thoracic/systemic diseases, drugs for sexual dysfunction (erectile dysfunction)

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 46 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF-5) | It will be measured after 12 weeks of training
  it will assess the sexual dysfunction in men

SECONDARY OUTCOMES:
alanine transaminase | It will be measured after 12 weeks of training
  it is an enzyme of liver will assess the liver funtions
aspartate transaminase | It will be measured after 12 weeks of training
  it is an enzyme of liver will assess the liver funtions
Rosenberg Self-Esteem Scale | It will be measured after 12 weeks of training
  it is a questionnaire that will assess Self-Esteem
Profile of Mood States | It will be measured after 12 weeks of training
  it is a questionnaire that will assess mood of men
depression inventory of Beck | It will be measured after 12 weeks of training
  it is a questionnaire that will assess depression of men

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt